CLINICAL TRIAL: NCT04441710
Title: Caregiver Serological Monitoring Extended Secondarily to Patients With the SARS-CoV-2 Coronavirus
Acronym: CoVid3S
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0395
Record Dates: First submitted 2020-06-18; First posted 2020-06-22 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: COVID
Keywords: COVID-19; SARS-COV-2; Serology; Predictability
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Caregivers: Staff of university hospitals
  Interventions: Other: Questionnaire
- Primary care caregivers: Population of professional caregivers such as general practitioner or freelance nurse.
  Interventions: Other: Questionnaire
- Patients
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Participants will be invited to complete a detailed questionnaire to collect prospectively and retrospectively data around the CoViD19 serological screening.

SUMMARY:
Hospital mortality attributed to SARS-CoV-2 in France increased daily by 28% in the week before confinement. The week following this decision, the daily increase was 30%. During the week of the second week of confinement, it started a decline of 19% estimated over the last 5 days, reaching the cumulative number of 2606 deaths on 29/3 (site https://www.eficiens.com/coronavirus- personal statistics / and calculation).

The diagnosis of viral carriage by RT-PCR is reserved for symptomatic cases among caregivers, due to the shortage of available tests and the cumbersome implementation. The carrier diagnosis is the benchmark, on which are implemented the therapeutic strategies and established the national statistics. It can present false negatives, linked to a research too early or too late in relation to the infection, or to a technical defect of the nasal swab sample. Caregivers on the front line in patient care, in hospitals or in the city, have only partial access to this diagnostic test, depending on the existence of symptoms. The implementation of a systematic serological screening, planned by the government and which cannot be based only on the search for the virus, will make it possible to inform the caregivers presenting symptoms or not, of their serological status, and therefore of their degree immunity or, on the contrary, susceptibility to infectious contacts. It should therefore be very voluntarily requested. On the occasion of this screening, the constitution of the COVID-3S cohort will make it possible to verify the degree of contamination in an asymptomatic population, information which is sorely lacking for the estimation of the immune coverage of the population. The implementation of the Covid-3S study will be based on the work of the National Reference Center of Pr B Lina, from the COVID-SER cohort, for the selection of the most efficient test (s). It seems useful to initiate the constitution of this cohort as soon as possible in relation to the evolution of the epidemic. Pending receipt of official recommendations, the lack of knowledge of the performance of serological tests means that it should be applied first to health professionals, better able to appreciate its limits, for the initial period before determining a validated serological screening strategy. Once the strategy has been specified, the gradual expansion of screening to the patient population will provide a more representative basis for the construction of epidemiological models for evaluating strategies.

ELIGIBILITY:
Inclusion Criteria:

* Any adult having passed a serological, antigenical or any other type of test in France, and voluntary to participate in the cohort and/or vaccinated against COVID19
* Any child under 18 who has passed a serological, antigenical, or any other type of test in France, willing to participate and at least one of whose parents has accepted to participate in the cohort, and/or vaccinated against COVID19

Exclusion Criteria:

* Persons deprived of their liberty
* Adults over whom legal protection applies: guardianship, curatorship

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Prospective cohort of voluntary caregivers, initially recruited in the CHUs concerned, then among the primary care caregivers, finally among the patients whom these caregivers care for.
Sampling Method: Non-Probability Sample
Enrollment: 2777 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Establishment of a reliable prediction model for the effectiveness of virus control | 18 months
  Estimated number of deaths avoided by the various population protection strategies, estimated by applying these strategies to the realistic virtual population.

CONTACTS AND LOCATIONS:
Overall Officials: Pascal FASCIA, MD, Principal Investigator — Hospices Civils de Lyon; François GUEYFFIER, MD, Study Director — Hospices Civils de Lyon
Locations (4):
- France (4):
  - CHU de Grenoble - Hôpital Nord, La Tronche
  - Hôpital de la Croix Rousse, Lyon
  - CHU de Saint Etienne, Saint-Etienne
  - Hôpital Henry Gabrielle, Saint-Genis-Laval